CLINICAL TRIAL: NCT00003111
Title: Phase II Clinical and Laboratory Study of Irinotecan/Cisplatin Chemotherapy Followed by Surgery in Stage III NSCLC
Brief Title: Combination Chemotherapy Followed by Surgery in Treating Patients With Stage IIIA Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065855; YALE-HIC-9317; NCI-G97-1345
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2009-08

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; Irinotecan; Paclitaxel; Neoadjuvant Therapy; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: irinotecan hydrochloride
Drug: paclitaxel
Procedure: neoadjuvant therapy
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with irinotecan and cisplatin followed by surgery in treating patients with stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of irinotecan based chemotherapy in patients with stage IIIA non-small cell lung cancer.
* Investigate the phenotypic changes induced in the tumor by this treatment.

OUTLINE: Patients receive IV cisplatin over 30 minutes followed by IV irinotecan over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for 3 courses until disease progression. Once potential candidates for resectability are determined, patients undergo thoracotomy or concurrent chemotherapy/radiation therapy within 6 weeks of completing the last course of chemotherapy. Following resection, patients responding to chemotherapy receive 3 additional courses of IV carboplatin and paclitaxel over 3 hours. Patients may undergo local irradiation beginning with the second course of carboplatin and paclitaxel. Chemotherapy ceases if disease remains stable after 8 weeks.

Patients are followed every 3 months for the first year after treatment, then every 6 months thereafter for survival.

PROJECTED ACCRUAL: This study will accrue 20 patients over 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed, previously untreated stage IIIa (T1-2 N2 M0) non-small cell lung cancer

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Total bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine clearance at least 55 mL/min

Other:

* Not HIV positive
* No active infections
* Not pregnant or lactating
* Effective contraception required of fertile patients during study participation
* No coexisting medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiation therapy
* No concurrent radiation therapy

Surgery:

* Not specified

Other:

* No concurrent use of investigational agents during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1997-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Murren, MD, Study Chair — Yale University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States